CLINICAL TRIAL: NCT03125655
Title: Regulation of Inflammatory Genes in Psoriasis
Status: Recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Nabiha Yusuf, Professor, University of Alabama at Birmingham
Other Study IDs: F120628003
Record Dates: First submitted 2017-04-17; First posted 2017-04-24 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-03

CONDITIONS: Psoriasis; Inflammation
Keywords: cytokines
MeSH Terms: conditions — Psoriasis; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Inflammatory markers

SUMMARY:
Psoriasis is a chronic and recurrent skin disorder characterized by marked inflammatory changes in the skin. An extensive cytokine network including generated by activated dendritic cells and T cells mediates the formation of psoriatic lesions. These immune-response parameters can be used as markers in the severity and management of the disease after further in-depth studies.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of psoriasis
* Must be age 19 or older.
* Must be Fitzpatrick skin type I, II, III, IV, V, VI.

Exclusion Criteria:

* Subjects who do not have photosensitive disease and are not on photosensitizing medications.
* Subjects with a history of keloids (who are more likely to develop hypertrophic scars following skin biopsy).
* Subjects who have an allergy to local anesthetics, antibiotics and/or anticoagulants.
* Subjects who are pregnant.

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects 19 and older will be recruited from the Dermatology clinics at UAB
Sampling Method: Probability Sample
Enrollment: 13 (Estimated)
Dates: Start 2014-04-22 (Actual); Primary Completion 2026-04-10 (Estimated); Study Completion 2027-04-28 (Estimated)

PRIMARY OUTCOMES:
Inflammatory genes | 1 day
  TNF-alpha , IFN-alpha , IL-6, IL-8, IL-12 , IL-23, IL-4, IL-5 and IL-10

CONTACTS AND LOCATIONS:
Locations (1):
- The Kirklin Clinic, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No